CLINICAL TRIAL: NCT02643732
Title: Fatigue in Sarcoidosis - A Feasibility Study Investigating the Treatment of Fatigue in Stable Sarcoidosis Patients Using Methylphenidate
Brief Title: Fatigue in Sarcoidosis - Treatment With Methylphenidate
Acronym: FaST-MP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of East Anglia (Other)
Collaborators: Clinical Research and Trials Unit (Norfolk & Norwich University Hospital, UK) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 170-11-15
Record Dates: First submitted 2015-12-23; First posted 2015-12-31 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Sarcoidosis; Fatigue
Keywords: Activity
MeSH Terms: conditions — Sarcoidosis; Fatigue; Motor Activity | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methylphenidate (Experimental): Methylphenidate 10mg (one tablet) twice daily, increasing to 20mg (two tablets) twice daily following assessment 2 weeks into trial.
  24 weeks duration
  Interventions: Drug: Methylphenidate (overencapsulated)
- Placebo (Placebo Comparator): Identical, over-encapsulated placebo tablets manufactured to be identical to the experimental tablets. One tablet twice daily, increased to two tablets twice daily following assessment 2 weeks into trial.
  24 weeks duration.
  Interventions: Drug: Placebo (Over-encapsulated tablet)

INTERVENTIONS:
Drug: Methylphenidate (overencapsulated) — 10mg (1 capsule) methylphenidate (standard release) twice daily, increased to 20mg (2 capsules) twice daily after 2 weeks. The drug can be down-titrated in the event of side effects, although re-uptitration is not allowed even if the side effects resolve on the lower dose.
  Other Names: Tranquilyn
  Arms: Methylphenidate
Drug: Placebo (Over-encapsulated tablet) — Identical capsules (over-encapsulated placebo tablets), administered initially one capsule twice daily, increased to 2 capsules after 2 weeks. As with the methylphenidate arm, the dose can be down-titrated in the event of side effects, although re-uptitration is not allowed even if the side effects resolve on the lower dose.
  Arms: Placebo

SUMMARY:
This is a small randomised-controlled trial (RCT) using methylphenidate as a treatment for clinically-significant fatigue in sarcoidosis patients with stable disease. The primary outcomes are feasibility, aimed at determining factors that will influence the design a future, larger RCT, which will be powered to look at clinical efficacy of the intervention.

DETAILED DESCRIPTION:
Sarcoidosis and fatigue

Sarcoidosis is a systemic granulomatous disease that affects all ethnic groups and ages. In the United Kingdom the incidence of the disease is 5.0 cases per 100,000 patient years, with a mean age at diagnosis of 47 years, frequently affecting patients of working age(Gribbin et al). The cause is unknown and there is no cure(Iannuzzi et al). Many patients suffer from debilitating fatigue for which there is presently no treatment.

Fatigue has been described as a "core symptom" of sarcoidosis, and is present in up to 80% of patients(Marcellis et al). A "post-sarcoidosis chronic-fatigue syndrome" has been described(James), denoting the presence of fatigue where there is no evidence of active disease. The presence of this symptom has been shown to adversely affect quality of life(Michielsen et al). Although there increased risk of obstructive sleep apnoea and sleep-disordered breathing occurring in sarcoidosis patients(Michielsen et al; Drent et al) the majority of patients have no identifiable cause for fatigue other than their sarcoidosis.

Both the British Thoracic Society(Bradley et al) and American Thoracic Society(Costabel et al) produce guidelines for physicians treating people with sarcoidosis. Neither guideline gives any advice on treatment of fatigue. Fatigue is a common problem in sarcoidosis. In a study of 76 patients with sarcoidosis, 50.7% reported pathological levels of fatigue, defined as a Fatigue Assessment Scale (FAS) score of greater than 21 units, compared with 8.6% of controls. People reporting fatigue scores above 21, had poorer EuroQoL Visual Analogue Scale (EQVAS) scores compared with people reporting fatigue scores of 21 or below (mean scores 0.561 vs 0.792 , p<0.001) (Unpublished data, Norfolk and Norwich University Hospital). This shows that fatigue impacts upon quality of life in sarcoidosis.

Methylphenidate - a treatment for fatigue

Methylphenidate (and its isomer dexmethylphenidate), which is used to treat attention deficit hyperactivity disorder(Keating et al), is an amphetamine-derivative which works by amplifying dopamine signals through inhibition of dopamine reuptake and enhancement of extracellular dopamine in the basal ganglia(Volkow et al). It has been used to treat fatigue in other settings with good effect. In a placebo-controlled, double-blind trial in post-chemotherapy participants with fatigue, methylphenidate exhibited a clinically significant reduction in fatigue(Lower et al). Prior to the results from this trial, a Cochrane review of treatments for cancer-related fatigue from 5 RCTs had shown an improvement in fatigue through methylphenidate treatment, leading them to conclude "the current evidence supports the use of psychostimulants in cancer-related fatigue"(Minton et al). Another trial investigated methylphenidate for the treatment of fatigue in 109 HIV-positive patients over a 6-week period. Methylphenidate improved fatigue on a visual analogue scale, with a 26.2 point increase (maximum of 100) from baseline, with 41% of participants receiving the drug demonstrating a greater than 50% improvement in visual analogue scale score(Breitbart et al). In contrast, no difference between methylphenidate and placebo was seen in a cohort of 68 fatigued patients who had received radiotherapy for brain tumours followed over a 12 week period(Butler et al).

In the case of sarcoidosis, so far only one small study has investigated the use of dexmethylphenidate for fatigue(Lower et al). Ten patients were included in this double blind crossover trial. Participants reported clinically and statistically significant improvements in fatigue measured by both the FAS and the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) score after 8 weeks of treatment, although no statistically significant improvement was seen in six minute walk distance (6MWD) compared with placebo. The drug was well tolerated; all participants completed the study and no significant increase in side effects was noted between the patients receiving placebo and dexmethylphenidate.

Rationale for current study

Prior to designing a definitive study, issues about the feasibility of undertaking a sufficiently large trial require to be resolved. Completed trials have only used methylphenidate for 8-12 weeks, so sustainability of effect, tolerability of medications over a long period and retention of participants within the trial are unknown. Whilst the use of medications such as methylphenidate may not be used on a continuous basis in the clinical setting, their use on a 6-12 month basis may not be unreasonable, hence the need to review the effect of the medication over a longer period. Furthermore, it is unclear how many people would be willing to participate in a longer trial , and how many potential participants would be suitable for enrolment using our present inclusion and exclusion criteria. For this reason, a feasibility trial is necessary before committing to a larger trial.

In addition, this trial will evaluate exercise and activity through both a modified shuttle walk test (MSWT) and accelerometer-measured change in activity levels. Although methylphenidate has not been shown to significantly improve 6MWD(Lower et al), a larger study using a more responsive test may be required to evaluate exercise capacity in this setting. This could be because as a self-paced test it is a sub-maximal exercise test - this has been shown to be the case in a study of interstitial lung disease (ILD) patients (including sarcoidosis) where peak oxygen uptake, carbon dioxide uptake and ventilation were all lower during 6MWD than on cardiopulmonary exercise testing(Holland et al). By not reaching their maximum exercise level this may make the test less responsive to change. This is particularly relevant given that the ILD cohort who did not reach maximal exercise or oxygen uptake during their 6MWD were likely to be much more limited in cardiopulmonary function than the cohort anticipated to be enrolled in a study of treatment of fatigue and therefore much more likely to get closer to their peak oxygen uptake during a 6MWD. Given that activity levels measured by accelerometers in people with sarcoidosis is related to fatigue (Korenromp et al), this trial will evaluate the feasibility of using them as an outcome measure in a clinical trial, including whether participants will wear the devices for long enough (i.e. 4 days out of 7, at least 10 hours per day) to get valid data for estimating daily activity levels.

Study Design

This is a parallel-arm RCT including 30 participants, randomised on a 1.5:1 basis in favour of the active treatment arm (18 participants will receive methylphenidate, 12 will receive placebo). The rationale of this trial is to determine the feasibility of designing and performing a sufficiently large RCT in the future looking for proof of clinical effect of methylphenidate in the treatment of sarcoidosis-associated fatigue. As a result, this study is not powered to detect a clinical difference in a clinical outcome, although these will be measured and analysed (the estimate of effect size will be used for future power calculations). Therefore the primary outcomes regard feasibility and safety, not treatment effect (see Outcome Measures section).

Participants will receive either methylphenidate or placebo for 24 weeks, with a further assessment performed 6 weeks after completion of the trial. They will be carefully monitored over the initial 6 weeks to ensure that they are stable on the drug - during this time they will be seen every 2 weeks (at 0,2,4 and 6 weeks). Following this period they will be seen less frequently (at 12 and 24 weeks, with postal questionnaires performed at 18 weeks) to detect sustainability of effect. Determining if treatment effect is sustained over the second half of the trial period will help to establish how long any future trial will need to be. Although each participant is required to attend frequent visits to the hospital, this trial has been designed in conjunction with sarcoidosis patients and ensures that participant safety is paramount.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy-proven diagnosis of sarcoidosis or diagnosis of sarcoidosis from interstitial lung disease multidisciplinary team meeting after review of radiological and clinical information
2. Stable disease (treatment unchanged for 6 weeks, without anticipation of treatment change during trial period)
3. FAS score greater than 21 units
4. Able to give informed consent
5. In patients on warfarin therapy - Willing to consent to increased frequency of monitoring

Exclusion Criteria:

1. Evidence of co-existing obstructive sleep apnoea. Patients screened with a "STOP-Bang" questionnaire (acronym taken from individual questions within the questionnaire itself) score of greater than 4 must undertake overnight oximetry; they are excluded if this shows a desaturation index of more than 15 events per hour on overnight oximetry.
2. Documented history of significant cardiac disease (including cardiac sarcoid) OR associated disease which would increase risk of underlying coronary artery disease (cerebrovascular disease, previous stroke or peripheral vascular disease). Definitively treated cardiac disease e.g. previous myocardial infarction treated with stents or coronary artery bypass grafting with no ongoing symptoms is permitted.
3. Hyperthyroidism evidenced by abnormal screening thyroid function tests (Thyroid stimulating hormone level outside normal range of 0.35 - 3.50 milliunits/litre (mU/L) or thyroxine (T4) outside normal range of 8 - 21 picomoles per litre (pmol/L)).
4. History of seizures, excluding febrile convulsions whilst an infant.
5. Abnormal electrocardiogram (ECG) with evidence of arrhythmia (except first degree heart block which has been stable for 3 months).
6. Concomitant therapy with the following drugs:

   * Tricyclic antidepressants
   * Monoamine oxidase inhibitors
   * Tramadol or buprenorphine
   * Levodopa
   * Haloperidol and atypical antipsychotics
7. Glaucoma or raised intra-ocular pressure for any reason.
8. Patients with established liver disease defined as Child-Pugh class B or C.
9. Documented medical history of psychiatric disorders (excluding depression)
10. History of drug-dependence or addiction at any time
11. Female participant who is pregnant, lactating or planning pregnancy during the course of the trial
12. Female patient of childbearing potential unable or unwilling to take two acceptable forms of contraception (see exclusions section)
13. Receiving an investigational drug or biological agent within 6 weeks (or 5 times the half-life if this is longer) prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-05 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate (Feasibility outcome) | Up to 18 months (recruitment period duration)
  How quickly the 30 participants are recruited to the study (relates to feasibility criteria regarding number of centres that are likely to be needed in a future, larger randomised controlled trial). Up to 18 months is allowed for recruitment, based on 2 years for trial to be run and 24 weeks for final patient to complete study.
Number of potential participants excluded (Feasibility outcome) | Up to 18 months (recruitment period duration)
  A record of the number of participants screened for inclusion will be kept, including whether they entered the trial or not, and if they were excluded, for what reason(s) they were excluded. This relates to number of centres likely to be required for a future trial. Up to 18 months is allowed for recruitment, based on 2 years for trial to be run and 24 weeks for final patient to complete study.
Number of participants dropping out/Participant retention rate (Feasibility outcome) | 24 weeks (trial duration)
  Number of participants withdrawing/dropping out of the study, including reasons where able; enables estimation of drop-out rates so that future studies can be appropriately sized, and also whether there are safety issues (side-effects necessitating withdrawals or patients not tolerating medications) that would suggest a future study is unnecessary.
Side-effect rate (Feasibility and Safety outcome) | 24 weeks (trial duration)
  Number of participants reporting side effects; what they are, severity and need for discontinuation of study drug all required.
  A likert scale measuring specific symptoms (palpitations, insomnia, headaches and chest pains) is also administered and these results will be recorded and presented to see if there are differences between the two groups.
  Participants also have an ECG at all study visits; any change in ECG will be recorded and the number of participants required to discontinue medications will be recorded.
Number of missed or unfilled assessments (Feasibility outcome) | 24 weeks (trial duration)
  Identifies whether appropriate data is being collected within the trial.
Number of accelerometers returned with valid data (Feasibility outcome) | 24 weeks (trial duration)
  Accelerometers are a novel outcome in this study. Their use in a trial of this nature has not been performed before. We wish to see how many participants return the accelerometer devices at the three time points in the trial, and how many of these have valid data on them; this is defined as 4 or more days of use with 10 or more hours or data. It is designed to see if it is feasible to use these devices as an outcome measure in future trials.

SECONDARY OUTCOMES:
Fatigue Assessment Scale (FAS) (Clinical outcome) | 0,2,4,6,12,18,14 and 30 weeks
  Change in FAS after 24 weeks, including sustainability of effect between 12 and 24 weeks (does clinical effect wane? would a future trial need to be as long?). The trial is not powered for looking for clinical difference (30 patients chosen to answer the primary feasibility questions), hence this is the secondary outcome. However, the estimate of effect size will enable power calculations for future studies to be more accurate.
  The FAS is measured at weeks 0,2,4,6,12,18,24 and 30 (6 weeks post-trial completion)
Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) | 0,2,4,6,12,18,14 and 30 weeks
  Change in FACIT-F after 24 weeks, including sustainability of effect - this question is co-administered with the FAS questionnaire, as performed in a small previous study (Lower EE et al, 2008).
  The FACIT-F is measured at weeks 0,2,4,6,12,18,24 and 30 (6 weeks post-trial completion)
Kings Sarcoidosis Questionnaire (KSQ) | 0,6,12,18,14 and 30 weeks
  The KSQ is a disease-specific, health-related quality of life score used in sarcoidosis and validated in sarcoidosis cohorts within the United Kingdom. It consists of 31 questions which require rating of health problems on a scale.
  The KSQ is assessed at weeks 0,6,12,18, 24 and 30 (6 weeks post-trial completion)
EuroQoL-5D (EQ5D) Questionnaire | 0,6,12,18,14 and 30 weeks
  This generic quality of life/health status questionnaire is used both to assess health status and also for exploratory health economic analysis.
  The EQ5D is performed at weeks 0,6,12,18,24 and 30 (6 weeks post-trial completion)
Short-form 36 (SF-36) Questionnaire | 0,6,12,18,14 and 30 weeks
  The SF-36 is a generic quality of life/health status questionnaire, which can also be used for health economic modelling. Both EQ5D and SF-36 are used here as the SF-36 has a vitality domain which can reflect changes in fatigue; the two questionnaires are therefore being compared to see which would be better to use in a future trial for both assessment of health status and health economic modelling.
  The SF-36 is performed at weeks 0,6,12,18,24 and 30 (6 weeks post-trial completion)
Hospital Anxiety and Depressions Score (HADS) | 0,6,12,18,14 and 30 weeks
  Depression has been suggested as a possible cause for fatigue in sarcoidosis, but it has also been suggested that the depression stems from the fatigue. Therefore a questionnaire identifying depressive and anxiety symptoms is administered.
  The HADS is performed at weeks 0,6,12,18,24 and 30 (6 weeks post-trial completion).
Accelerometer Use (wrist-worn accelerometer) | 0, 12, 24 weeks
  A wrist-worn accelerometer can measure daily activity levels over a 7 day period. This will be performed before commencing medication (between screening and baseline visit), at the mid-point (12 weeks) and in the 2 weeks prior to medication completion (22-24 weeks). This will enable assessment in change of activity levels between the groups.
Modified Shuttle Walk Test (MSWT) | 0, 12, 24 weeks
  This incremental physical exercise test will enable an assessment in change in physical capacity/ability to be made. Like the accelerometer outcome, it is assessed at 0,12 and 24 weeks.

OTHER OUTCOMES:
Health Economic/Utility Use | 0, 12, 24 weeks
  A custom questionnaire based on existing tools will be administered at weeks 0,12 and 24 to look for changes in use of health and social facilities/services, as well as time off work/change in working patterns.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M Wilson, MD, Principal Investigator — University of East Anglia
Locations (1):
- Norfolk and Norwich University Hospital, Norwich, Norfolk, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Plan for anonymised data to be available through data repository for analysis by other researchers with permission of team.

REFERENCES:
- [Background] Gribbin J, Hubbard RB, Le Jeune I, Smith CJ, West J, Tata LJ. Incidence and mortality of idiopathic pulmonary fibrosis and sarcoidosis in the UK. Thorax. 2006 Nov;61(11):980-5. doi: 10.1136/thx.2006.062836. Epub 2006 Jul 14. PMID 16844727
- [Background] Iannuzzi MC, Rybicki BA, Teirstein AS. Sarcoidosis. N Engl J Med. 2007 Nov 22;357(21):2153-65. doi: 10.1056/NEJMra071714. No abstract available. PMID 18032765
- [Background] Marcellis RG, Lenssen AF, Elfferich MD, De Vries J, Kassim S, Foerster K, Drent M. Exercise capacity, muscle strength and fatigue in sarcoidosis. Eur Respir J. 2011 Sep;38(3):628-34. doi: 10.1183/09031936.00117710. Epub 2011 Mar 24. PMID 21436356
- [Background] James DG. Complications of sarcoidosis. Chronic fatigue syndrome. Sarcoidosis. 1993 Mar;10(1):1-3. PMID 8134708
- [Background] Michielsen HJ, Drent M, Peros-Golubicic T, De Vries J. Fatigue is associated with quality of life in sarcoidosis patients. Chest. 2006 Oct;130(4):989-94. doi: 10.1378/chest.130.4.989. PMID 17035429
- [Background] Turner GA, Lower EE, Corser BC, Gunther KL, Baughman RP. Sleep apnea in sarcoidosis. Sarcoidosis Vasc Diffuse Lung Dis. 1997 Mar;14(1):61-4. PMID 9186990
- [Background] Drent M, Verbraecken J, van der Grinten C, Wouters E. Fatigue associated with obstructive sleep apnea in a patient with sarcoidosis. Respiration. 2000;67(3):337-40. doi: 10.1159/000029523. PMID 10867608
- [Background] Bradley B, Branley HM, Egan JJ, Greaves MS, Hansell DM, Harrison NK, Hirani N, Hubbard R, Lake F, Millar AB, Wallace WA, Wells AU, Whyte MK, Wilsher ML; British Thoracic Society Interstitial Lung Disease Guideline Group, British Thoracic Society Standards of Care Committee; Thoracic Society of Australia; New Zealand Thoracic Society; Irish Thoracic Society. Interstitial lung disease guideline: the British Thoracic Society in collaboration with the Thoracic Society of Australia and New Zealand and the Irish Thoracic Society. Thorax. 2008 Sep;63 Suppl 5:v1-58. doi: 10.1136/thx.2008.101691. No abstract available. PMID 18757459
- [Background] Costabel U, Hunninghake GW. ATS/ERS/WASOG statement on sarcoidosis. Sarcoidosis Statement Committee. American Thoracic Society. European Respiratory Society. World Association for Sarcoidosis and Other Granulomatous Disorders. Eur Respir J. 1999 Oct;14(4):735-7. doi: 10.1034/j.1399-3003.1999.14d02.x. No abstract available. PMID 10573213
- [Background] Keating GM, Figgitt DP. Dexmethylphenidate. Drugs. 2002;62(13):1899-904; discussion 1905-8. doi: 10.2165/00003495-200262130-00009. PMID 12215063
- [Background] Volkow ND, Fowler JS, Wang G, Ding Y, Gatley SJ. Mechanism of action of methylphenidate: insights from PET imaging studies. J Atten Disord. 2002;6 Suppl 1:S31-43. doi: 10.1177/070674370200601s05. PMID 12685517
- [Background] Lower EE, Fleishman S, Cooper A, Zeldis J, Faleck H, Yu Z, Manning D. Efficacy of dexmethylphenidate for the treatment of fatigue after cancer chemotherapy: a randomized clinical trial. J Pain Symptom Manage. 2009 Nov;38(5):650-62. doi: 10.1016/j.jpainsymman.2009.03.011. PMID 19896571
- [Background] Minton O, Richardson A, Sharpe M, Hotopf M, Stone P. Drug therapy for the management of cancer-related fatigue. Cochrane Database Syst Rev. 2010 Jul 7;2010(7):CD006704. doi: 10.1002/14651858.CD006704.pub3. PMID 20614448
- [Background] Breitbart W, Rosenfeld B, Kaim M, Funesti-Esch J. A randomized, double-blind, placebo-controlled trial of psychostimulants for the treatment of fatigue in ambulatory patients with human immunodeficiency virus disease. Arch Intern Med. 2001 Feb 12;161(3):411-20. doi: 10.1001/archinte.161.3.411. PMID 11176767
- [Background] Butler JM Jr, Case LD, Atkins J, Frizzell B, Sanders G, Griffin P, Lesser G, McMullen K, McQuellon R, Naughton M, Rapp S, Stieber V, Shaw EG. A phase III, double-blind, placebo-controlled prospective randomized clinical trial of d-threo-methylphenidate HCl in brain tumor patients receiving radiation therapy. Int J Radiat Oncol Biol Phys. 2007 Dec 1;69(5):1496-501. doi: 10.1016/j.ijrobp.2007.05.076. Epub 2007 Sep 14. PMID 17869448
- [Background] Lower EE, Harman S, Baughman RP. Double-blind, randomized trial of dexmethylphenidate hydrochloride for the treatment of sarcoidosis-associated fatigue. Chest. 2008 May;133(5):1189-95. doi: 10.1378/chest.07-2952. Epub 2008 Feb 8. PMID 18263672
- [Background] Holland AE, Dowman L, Fiore J Jr, Brazzale D, Hill CJ, McDonald CF. Cardiorespiratory responses to 6-minute walk test in interstitial lung disease: not always a submaximal test. BMC Pulm Med. 2014 Aug 11;14:136. doi: 10.1186/1471-2466-14-136. PMID 25113781
- [Background] Korenromp IHE, Heijnen CJ, Vogels OJM, van den Bosch JMM, Grutters JC. Characterization of chronic fatigue in patients with sarcoidosis in clinical remission. Chest. 2011 Aug;140(2):441-447. doi: 10.1378/chest.10-2629. Epub 2011 Feb 17. PMID 21330380
- [Derived] Atkins C, Jones A, Clark AB, Stockl A, Fordham R, Wilson AM. Feasibility of investigating methylphenidate for the treatment of sarcoidosis-associated fatigue (the FaST-MP study): a double-blind, parallel-arm randomised feasibility trial. BMJ Open Respir Res. 2021 May;8(1):e000814. doi: 10.1136/bmjresp-2020-000814. PMID 34020962
- [Derived] Atkins C, Fordham R, Clark AB, Stockl A, Jones AP, Wilson AM. Feasibility study of a randomised controlled trial to investigate the treatment of sarcoidosis-associated fatigue with methylphenidate (FaST-MP): a study protocol. BMJ Open. 2017 Dec 4;7(12):e018532. doi: 10.1136/bmjopen-2017-018532. PMID 29208618